CLINICAL TRIAL: NCT00846586
Title: A Randomized, Double-blind, Controlled, Parallel-group, 12-week Study to Compare the Efficacy and Safety of the Combination of Indacaterol 150 µg Once Daily With Open Label Tiotropium 18 µg Once Daily Versus Open Label Tiotropium 18 µg Once Daily in Patients With Moderate-to-severe Chronic Obstructive Pulmonary Disease
Brief Title: Efficacy and Safety of Indacaterol Plus Tiotropium Versus Tiotropium Alone in Patients With Chronic Obstructive Pulmonary Disease
Acronym: INTRUST1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149B2341
Record Dates: First submitted 2009-02-15; First posted 2009-02-18 (Estimated); Results first posted 2011-08-18 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: chronic obstructive pulmonary disease; COPD; indacaterol; tiotropium; bronchodilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Indacaterol 150 μg and tiotropium 18 μg (Experimental): Patients inhaled indacaterol 150 μg and tiotropium 18 μg once daily in the morning between 8:00 AM and 11:00 AM for 12 weeks. Indacaterol was delivered blinded via a single dose dry powder inhaler (SDDPI). Tiotropium was delivered open-label via the manufacturer's proprietary inhalation device (HandiHaler®). Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 150 μg; Drug: Tiotropium 18 μg
- Tiotropium 18 μg (Active Comparator): Patients inhaled placebo to indacaterol 150 μg and tiotropium 18 μg once daily in the morning between 8:00 AM and 11:00 AM for 12 weeks. Placebo to indacaterol was delivered blinded via a single dose dry powder inhaler (SDDPI). Tiotropium was delivered open-label via the manufacturer's proprietary inhalation device (HandiHaler®). Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Tiotropium 18 μg; Drug: Placebo to indacaterol

INTERVENTIONS:
Drug: Indacaterol 150 μg — Indacaterol was supplied in powder filled capsules together with a single dose dry powder inhaler (SDDPI) device.
  Arms: Indacaterol 150 μg and tiotropium 18 μg
Drug: Tiotropium 18 μg — Tiotropium was supplied in powder filled capsules together the manufacture's proprietary inhalation device (HandiHaler®).
Drug: Placebo to indacaterol — Placebo to indacaterol was supplied in powder filled capsules together with a single dose dry powder inhaler (SDDPI) device.
  Arms: Tiotropium 18 μg

SUMMARY:
This study assessed the efficacy and safety of indacaterol (150 µg once daily [od]) when combined with tiotropium (18 µg od) versus tiotropium (18 µg od) treatment alone in patients with chronic obstructive pulmonary disease (COPD)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic obstructive pulmonary disease (COPD) (moderate-to-severe as classified by the Global Initiative for Chronic Obstructive Lung Disease [GOLD] Guidelines, 2007) and:

  1. Smoking history of at least 10 pack-years
  2. Post-bronchodilator forced expiratory volume in 1 second (FEV1) ≤ 65% and ≥ 30% of the predicted normal value
  3. Post-bronchodilator FEV1/FVC (force vital capacity) < 70%

Exclusion Criteria:

* Patients who have had a COPD exacerbation requiring systemic glucocorticosteroid treatment or antibiotics and/or hospitalization in the 6 weeks prior to screening or during the run-in period
* Patients who have had a respiratory tract infection within 6 weeks prior to screening or during the run-in period
* Patients with a body mass index less than 15 or more than 40 kg/m^2
* Patients with concomitant pulmonary disease
* Patients with a history of asthma
* Patients with diabetes Type I or uncontrolled diabetes Type II
* Any patient with lung cancer or a history of lung cancer
* Patients with a history of certain cardiovascular comorbid conditions

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1134 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (134):
- United States (58):
  - Novartis Investigator Site, Birmingham, Alabama
  - Novartis Investigator Site, Mobile, Alabama
  - Novartis Investigative Site, Scottsdale, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigator Site, Pine Bluff, Arkansas
  - Novartis Investigator Site, Fountain Valley, California
  - Novartis Investigator Site, Long Beach, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigator Site, National City, California
  - Novartis Investigator Site, Palmdale, California
  - Novartis Investigative Site, Stockton, California
  - Novartis Investigator Site, Temecula, California
  - Novartis Investigative Site, Hartford, Connecticut
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigator Site, Fort Walton Beach, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Naranja, Florida
  - Novartis Investigator Site, Pensacola, Florida
  - Novartis Investigator Site, Sarasota, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigator Site, Conyers, Georgia
  - Novartis Investigative Site, Normal, Illinois
  - Novartis Investigative Site, Iowa City, Iowa
  - Novartis Investigative Site, Kansas City, Kansas
  - Novartis Investigative Site, Lenexa, Kansas
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigator Site, Lafayette, Louisiana
  - Novartis Investigator Site, Metaire, Louisiana
  - Novartis Investigator Site, New Orleans, Louisiana
  - Novartis Investigator Site, Slidell, Louisiana
  - Novartis Investigator Site, Columbia, Maryland
  - Novartis Investigator Site, Brockton, Massachusetts
  - Novartis Investigator Site, Clarkston, Michigan
  - Novartis Investigator Site, Detroit, Michigan
  - Novartis Investigative Site, Saint Charles, Missouri
  - Novartis Investigator Site, Missoula, Montana
  - Novartis Investigator Site, Boys Town, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative site, Omaha, Nebraska
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigator Site, Lebanon, New Hampshire
  - Novartis Investigator Site, Asbury Park, New Jersey
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigator Site, Mooresville, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigator Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigator Site, Bethlehem, Pennsylvania
  - Novartis Investigative Site, Cumberland, Rhode Island
  - Novartis Investigator Site, Greenville, South Carolina
  - Novartis Investigative Site, Spartanburg, South Carolina
  - Novartis Investigator Site, Knoxville, Tennessee
  - Novartis Investigator Site, El Paso, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Center, New Braunfels, Texas
  - Novartis Investigator Site, Newport News, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigator Site, Richmond, Virginia
- Argentina (5):
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Corrientes
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative SIte, Mendoza
  - Novartis Investigative Site, Rosario
- Australia (6):
  - Novartis Investigator Site, Box Hill
  - Novartis Investigator Site, Clayton
  - Novartis Investigator Site, Garran
  - Novartis Investigator Site, Glebe
  - Novartis Investigator Site, Kogarah
  - Novartis Investigator Site, Nedlands
- Colombia (4):
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Bogotá
  - Novartis Investigator Site, Bogotá
  - Novartis Investigative Site, Medellín
- Denmark (5):
  - Novartis Investigator Site, Copenhagen
  - Novartis Investigator Site, Fredericia
  - Novartis Investigator Site, Silkeborg
  - Novartis Investigator Site, Soeborg
  - Novartis Investigator Site, Vejle
- Germany (21):
  - Novartis Investigator Site, Berlin
  - Novartis Investigator Site, Cottbus
  - Novartis Investigator Site, Donaustauf
  - Novartis Investigator Site, Dortmund
  - Novartis Investigator Site, Erfurt
  - Novartis Investigator Site, Frankfurt
  - Novartis Investigator Site, Gelnhausen
  - Novartis Investigator Site, Großhansdorf
  - Novartis Investigator Site, Hanover
  - Novartis Investigator Site, Heidelberg
  - Novartis Investigator Site, Leipzig
  - Novartis Investigator Site, Mainz
  - Novartis Investigator Site, Neu-Ulm
  - Novartis Investigator Site, Neuss
  - Novartis Investigator Site, Potsdam
  - Novartis Investigator Site, Rostock
  - Novartis Investigator Site, Schwabach
  - Novartis Investigator Site, Schwetzingen
  - Novartis Investigator Site, Straußberg
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigator Site, Wuppertal
- Novartis Investigative Site, Guatemala City, Guatemala
- Mexico (4):
  - Novartis Investigative Site, Guadalajara
  - Novartis Investigator Site, Mexico City
  - Novartis Investigative Site, Monterrey
  - Novartis Investigative Site, Zapopan
- Novartis Investigator Site, Manila, Philippines
- South Africa (5):
  - Novartis Investigator Site, Cape Town
  - Novartis Investigator Site, eManzimtoti
  - Novartis Investigator Site, eMkhomazi
  - Novartis Investigator Site, Johannesburg
  - Novartis Investigator Site, Midrand
- Spain (13):
  - Novartis Investigator Site, A Coruña
  - Novartis Investigative Site, Alicante
  - Novartis Investigator Site, Barcelona
  - Novartis Investigator Site, Begonte
  - Novartis Investigator Site, Cadiz
  - Novartis Investigator Site, Granollers
  - Novartis Investigative Site, Jaén
  - Novartis Investigator Site, León
  - Novartis Investigator Site, Madrid
  - Novartis Investigator Site, Pamplona
  - Novartis Investigator Site, Torrelavega
  - Novartis Investigator Site, Valencia
  - Novartis Investigator Site, Vigo
- Turkey (Türkiye) (11):
  - Novartis Investigator Site, Antalya
  - Novartis Investigator Site, Çanakkale
  - Novartis Investigator Site, Isparta
  - Novartis Investigator Site, Istanbul
  - Novartis Investigator Site, Kartal
  - Novartis Investigator Site, Kayseri
  - Novartis Investigator Site, Kozlu / Zonguldak
  - Novartis Investigator Site, Malatya
  - Novartis Investigator Site, Manisa
  - Novartis Investigator Site, Mecidiyekoy/Istanbul
  - Novartis Investigator Site, Yenisehir/Izmir

REFERENCES:
- [Derived] Mahler DA, D'Urzo A, Bateman ED, Ozkan SA, White T, Peckitt C, Lassen C, Kramer B; INTRUST-1 and INTRUST-2 study investigators. Concurrent use of indacaterol plus tiotropium in patients with COPD provides superior bronchodilation compared with tiotropium alone: a randomised, double-blind comparison. Thorax. 2012 Sep;67(9):781-8. doi: 10.1136/thoraxjnl-2011-201140. Epub 2012 Apr 27. PMID 22544891

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Indacaterol 150 μg and Tiotropium 18 μg | Tiotropium 18 μg
Started | 570 | 564
Received Study Drug | 570 | 561 (Three patients were not exposed to study treatment in this group.)
Completed | 531 | 529
Not Completed | 39 | 35
Not completed — Adverse Event | 20 | 10
Not completed — Subject withdrew consent | 8 | 10
Not completed — Administrative problems | 5 | 4
Not completed — Death | 2 | 0
Not completed — Protocol deviation | 2 | 6
Not completed — Abnormal test procedure result(s) | 1 | 0
Not completed — Lost to Follow-up | 1 | 4
Not completed — Unsatisfactory therapeutic effect | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol 150 μg and Tiotropium 18 μg | Tiotropium 18 μg | Total
Number analyzed (Participants) | 570 | 561 | 1131
Age Continuous [Mean (Standard Deviation); unit: years] — Demographics are reported for the safety set which includes all patients who received at least 1 dose of study drug.
  years | 64.0 (9.07) | 63.4 (9.22) | 63.7 (9.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171 | 183 | 354
  Male | 399 | 378 | 777

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Standardized (With Respect to Length of Time) Area Under the Curve (AUC) From 5 Minutes to 8 Hours Post-dose at the End of Treatment (Week 12)
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made at 5 and 30 minutes; and 1, 2, 3, 4, 6, and 8 hours post-dose at the end of the study (Week 12, Day 84). Standardized FEV1 AUC was calculated by the trapezoidal rule. The analysis included baseline FEV1, FEV1 pre-dose and 10-15 minutes post-dose of salbutamol/albuterol during screening, and FEV1 pre-dose and 1 hour post-dose of ipratropium during screening as covariates.
Time Frame: From 5 minutes to 8 hours post-dose at the end of treatment (Week 12, Day 84)
Population: Full analysis set (FAS): All randomized patients who received at least 1 dose of study drug, last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg and Tiotropium 18 μg | Tiotropium 18 μg
Number analyzed (Participants) | 505 | 504
Liters | 1.50 (0.014) | 1.38 (0.014)

2. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) 24 Hours Post-dose at the End of Treatment (Week 12 + 1 Day, Day 85)
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made at 23 hours 10 minutes and 23 hours 45 minutes post-dose at the end of the study (Week 12 + 1 day, Day 85). The analysis included baseline FEV1, FEV1 pre-dose and 10-15 minutes post-dose of salbutamol/albuterol during screening, and FEV1 pre-dose and 1 hour post-dose of ipratropium during screening as covariates.
Time Frame: 24 hours post-dose at the end of treatment (Week 12 + 1 day, Day 85)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg and Tiotropium 18 μg | Tiotropium 18 μg
Number analyzed (Participants) | 561 | 549
Liters | 1.38 (0.014) | 1.30 (0.014)

3. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Standardized (With Respect to Length of Time) Area Under the Curve (AUC) From 5 Minutes to 8 Hours Post-dose on Day 1
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made at 5 and 30 minutes; and 1, 2, 3, 4, 6, and 8 hours post-dose on Day 1. Standardized FEV1 AUC was calculated by the trapezoidal rule. The analysis included baseline FEV1, FEV1 pre-dose and 10-15 minutes post-dose of salbutamol/albuterol during screening, and FEV1 pre-dose and 1 hour post-dose of ipratropium during screening as covariates.
Time Frame: From 5 minutes to 8 hours post-dose on Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg and Tiotropium 18 μg | Tiotropium 18 μg
Number analyzed (Participants) | 544 | 523
Liters | 1.40 (0.009) | 1.32 (0.009)

4. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) 24 Hours Post-dose on Day 2
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made at 23 hours 10 minutes and 23 hours 45 minutes post-dose on Day 2. The analysis included baseline FEV1, FEV1 pre-dose and 10-15 minutes post-dose of salbutamol/albuterol during screening, and FEV1 pre-dose and 1 hour post-dose of ipratropium during screening as covariates.
Time Frame: 24 hours post-dose on Day 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg and Tiotropium 18 μg | Tiotropium 18 μg
Number analyzed (Participants) | 553 | 541
Liters | 1.36 (0.011) | 1.27 (0.012)

5. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Standardized (With Respect to Length of Time) Area Under the Curve (AUC) From 5 Minutes to 4 Hours Post-dose on Day 1
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made at 5 and 30 minutes; and 1, 2, 3, and 4 hours post-dose on Day 1. Standardized FEV1 AUC was calculated by the trapezoidal rule. The analysis included baseline FEV1, FEV1 pre-dose and 10-15 minutes post-dose of salbutamol/albuterol during screening, and FEV1 pre-dose and 1 hour post-dose of ipratropium during screening as covariates.
Time Frame: From 5 minutes to 4 hours post-dose on Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg and Tiotropium 18 μg | Tiotropium 18 μg
Number analyzed (Participants) | 552 | 527
Liters | 1.38 (0.008) | 1.31 (0.008)

6. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Standardized (With Respect to Length of Time) Area Under the Curve (AUC) From 5 Minutes to 4 Hours Post-dose at the End of Treatment (Week 12)
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made at 5 and 30 minutes; and 1, 2, 3, and 4 hours post-dose at the end of treatment (Week 12). Standardized FEV1 AUC was calculated by the trapezoidal rule. The analysis included baseline FEV1, FEV1 pre-dose and 10-15 minutes post-dose of salbutamol/albuterol during screening, and FEV1 pre-dose and 1 hour post-dose of ipratropium during screening as covariates.
Time Frame: From 5 minutes to 4 hours post-dose at the end of treatment (Week 12)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg and Tiotropium 18 μg | Tiotropium 18 μg
Number analyzed (Participants) | 516 | 511
Liters | 1.52 (0.013) | 1.38 (0.013)

ADVERSE EVENTS:
Time Frame: Baseline to the end of the study (Week 12)
Description: Safety set: All patients who received at least 1 dose of study drug.
Arm/Group | Indacaterol 150 μg and Tiotropium 18 μg | Tiotropium 18 μg
Serious Adverse Events (participants affected / at risk) | 21/570 | 17/561
Other Adverse Events (participants affected / at risk) | 99/570 | 69/561
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 μg and Tiotropium 18 μg (N=570) | Tiotropium 18 μg (N=561)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 2 | 0
Atrial flutter (Cardiac disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection bacterial (Infections and infestations) | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Bladder neck obstruction (Renal and urinary disorders) | 1 | 0
Myoglobinuria (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1
Residual urine (Renal and urinary disorders) | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Urine flow decreased (Renal and urinary disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Arterial disorder (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 μg and Tiotropium 18 μg (N=570) | Tiotropium 18 μg (N=561)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 48 | 51
Cough (Respiratory, thoracic and mediastinal disorders) | 59 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.